CLINICAL TRIAL: NCT04625283
Title: The Effect and Contribution of a Perioperative Ketamine Infusion in an Established Enhanced Recovery Pathway
Brief Title: The Impact of Perioperative Ketamine Infusion on Surgical Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Britany Lynn Raymond, MD, MD, Assistant Professor, Department of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200210
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Opioid Use; Enhanced Recovery After Surgery; Anesthesia; Ketamine; Pain, Postoperative
Keywords: ERAS; Enhanced Recovery After Surgery; Ketamine; Opioid; Learning Healthcare System
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study will be performed as a pragmatic controlled clinical trial with parallel group assignment. Randomization will be in a cluster format.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participants in this arm will receive intraoperative ketamine bolus (0.5mg/kg) followed by continuous infusion 5 mcg/kg/min and also will receive postoperative ketamine infusion (2.5 mcg/kg/min, up to 100kg max) for 48 hours.
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): Participants in this arm will receive an equivalent volume of intraoperative saline bolus followed by continuous saline infusion and also will receive postoperative saline infusion for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Participants in the ketamine arm will receive intraoperative and postoperative ketamine.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Placebo — Participants in the placebo arm will receive intraoperative and postoperative saline.
  Other Names: Saline
  Arms: Saline

SUMMARY:
In order to effectively treat surgical pain with the least amount of opioids required, a multi-modal approach must include medications with different mechanisms of actions at alternative receptors. In light of the opioid epidemic, medical providers at Vanderbilt University Medical Center (VUMC) are strategically combining these medications in a bundled pain-regimen after surgery. These regimens have been shown to decrease opioid consumption, improve surgical outcomes, and reduce hospital stays, thus coining the term 'enhanced recovery pathway'. The combination of these medications has an indisputable synergistic effect. However, it is unknown how each medication contributes individually to the overall efficacy of the pathway. This study will examine the effects of ketamine, within the constructs of a multimodal pain regimen, on a) length of stay, b) opioid consumption, and c) surgical outcomes after major abdominal surgery.

DETAILED DESCRIPTION:
Opioids are powerful analgesic medications that can reduce pain through action at the mu receptor. Unfortunately, activation of the mu receptor also results in undesirable side effects, such as respiratory depression, sedation, bowel ileus, nausea, itching, and tolerance. Therefore, in order to effectively treat pain with the least amount of opioids required, a multi-modal approach must include medications with different mechanisms of actions at alternative receptors. Some examples of non-narcotic pain medications include acetaminophen (Tylenol), anti-inflammatories (NSAIDS), muscle relaxants, local anesthetics, gabapentinoids (Lyrica), and ketamine, to name a few. In light of the opioid epidemic, medical providers at Vanderbilt University Medical Center (VUMC) are strategically combining these medications in a bundled pain-regimen after surgery. These regimens have been shown to decrease opioid consumption, improve surgical outcomes, and reduce hospital stays, thus coining the term 'enhanced recovery pathway' or enhanced recovery after surgery (ERAS). The combination of these medications has an indisputable synergistic effect. However, it is unknown how each medication contributes individually to the overall efficacy of the pathway. Ultimately, the investigators aim to perform a series of randomized controlled trials in which we isolate each component of the pathway to investigate its effects on length of stay, total opioid consumption, and surgical outcomes. The investigators will begin with studying ketamine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater
* presenting at VUMC for abdominal surgery on the colorectal, ventral hernia or surgical oncology services on a weekday.

Exclusion Criteria:

* allergy or contraindication to ketamine
* unable or refuse to receive a neuraxial or regional nerve block
* patient refusal
* direct transfer from operating room to intensive care unit with endotracheal tube placed
* treating team elects to exclude the patient prior to study drug administration
* abortion of planned surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1570 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britany L Raymond, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data.

REFERENCES:
- [Background] Boenigk K, Echevarria GC, Nisimov E, von Bergen Granell AE, Cuff GE, Wang J, Atchabahian A. Low-dose ketamine infusion reduces postoperative hydromorphone requirements in opioid-tolerant patients following spinal fusion: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jan;36(1):8-15. doi: 10.1097/EJA.0000000000000877. PMID 30113350
- [Background] Kaur S, Saroa R, Aggarwal S. Effect of intraoperative infusion of low-dose ketamine on management of postoperative analgesia. J Nat Sci Biol Med. 2015 Jul-Dec;6(2):378-82. doi: 10.4103/0976-9668.160012. PMID 26283834
- [Background] Kim SH, Kim SI, Ok SY, Park SY, Kim MG, Lee SJ, Noh JI, Chun HR, Suh H. Opioid sparing effect of low dose ketamine in patients with intravenous patient-controlled analgesia using fentanyl after lumbar spinal fusion surgery. Korean J Anesthesiol. 2013 Jun;64(6):524-8. doi: 10.4097/kjae.2013.64.6.524. Epub 2013 Jun 24. PMID 23814653
- [Background] Suppa E, Valente A, Catarci S, Zanfini BA, Draisci G. A study of low-dose S-ketamine infusion as "preventive" pain treatment for cesarean section with spinal anesthesia: benefits and side effects. Minerva Anestesiol. 2012 Jul;78(7):774-81. Epub 2012 Feb 29. PMID 22374377
- [Background] Remerand F, Le Tendre C, Baud A, Couvret C, Pourrat X, Favard L, Laffon M, Fusciardi J. The early and delayed analgesic effects of ketamine after total hip arthroplasty: a prospective, randomized, controlled, double-blind study. Anesth Analg. 2009 Dec;109(6):1963-71. doi: 10.1213/ANE.0b013e3181bdc8a0. PMID 19923527
- [Background] Pergolizzi JV Jr, Rosenblatt M, LeQuang JA. Three Years Down the Road: The Aftermath of the CDC Guideline for Prescribing Opioids for Chronic Pain. Adv Ther. 2019 Jun;36(6):1235-1240. doi: 10.1007/s12325-019-00954-1. Epub 2019 Apr 23. PMID 31016474
- [Background] Kent ML, Hurley RW, Oderda GM, Gordon DB, Sun E, Mythen M, Miller TE, Shaw AD, Gan TJ, Thacker JKM, McEvoy MD; POQI-4 Working Group. American Society for Enhanced Recovery and Perioperative Quality Initiative-4 Joint Consensus Statement on Persistent Postoperative Opioid Use: Definition, Incidence, Risk Factors, and Health Care System Initiatives. Anesth Analg. 2019 Aug;129(2):543-552. doi: 10.1213/ANE.0000000000003941. PMID 30897590
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Kurokawa Y, Kurokawa T, Tanimoto T. Opioid Prescription After Surgery. JAMA Surg. 2019 Jul 1;154(7):675. doi: 10.1001/jamasurg.2019.0573. No abstract available. PMID 31017640
- [Background] Mercadante S. Opioid Analgesics Adverse Effects: The Other Side of the Coin. Curr Pharm Des. 2019;25(30):3197-3202. doi: 10.2174/1381612825666190717152226. PMID 31333113
- [Background] McEvoy MD, Wanderer JP, King AB, Geiger TM, Tiwari V, Terekhov M, Ehrenfeld JM, Furman WR, Lee LA, Sandberg WS. A perioperative consult service results in reduction in cost and length of stay for colorectal surgical patients: evidence from a healthcare redesign project. Perioper Med (Lond). 2016 Feb 5;5:3. doi: 10.1186/s13741-016-0028-1. eCollection 2016. PMID 26855773
- [Background] Hawkins AT, Geiger TM, King AB, Wanderer JP, Tiwari V, Muldoon RL, Ford MM, Dmochowski RR, Sandberg WS, Martin B, Hopkins MB, McEvoy MD. An enhanced recovery program in colorectal surgery is associated with decreased organ level rates of complications: a difference-in-differences analysis. Surg Endosc. 2019 Jul;33(7):2222-2230. doi: 10.1007/s00464-018-6508-2. Epub 2018 Oct 17. PMID 30334161
- [Background] King AB, Spann MD, Jablonski P, Wanderer JP, Sandberg WS, McEvoy MD. An enhanced recovery program for bariatric surgical patients significantly reduces perioperative opioid consumption and postoperative nausea. Surg Obes Relat Dis. 2018 Jun;14(6):849-856. doi: 10.1016/j.soard.2018.02.010. Epub 2018 Feb 13. PMID 29555468
- [Background] Li Z, Zhao Q, Bai B, Ji G, Liu Y. Enhanced Recovery After Surgery Programs for Laparoscopic Abdominal Surgery: A Systematic Review and Meta-analysis. World J Surg. 2018 Nov;42(11):3463-3473. doi: 10.1007/s00268-018-4656-0. PMID 29750324
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Doan LV, Wang J. An Update on the Basic and Clinical Science of Ketamine Analgesia. Clin J Pain. 2018 Nov;34(11):1077-1088. doi: 10.1097/AJP.0000000000000635. PMID 29927768
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Peyton PJ, Wu C, Jacobson T, Hogg M, Zia F, Leslie K. The effect of a perioperative ketamine infusion on the incidence of chronic postsurgical pain-a pilot study. Anaesth Intensive Care. 2017 Jul;45(4):459-465. doi: 10.1177/0310057X1704500408. PMID 28673215
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Allen CA, Ivester JR Jr. Low-Dose Ketamine for Postoperative Pain Management. J Perianesth Nurs. 2018 Aug;33(4):389-398. doi: 10.1016/j.jopan.2016.12.009. Epub 2017 Jun 10. PMID 30077280
- [Background] Plyler SS, Muckler VC, Titch JF, Gupta DK, Rice AN. Low-Dose Ketamine Infusion to Decrease Postoperative Delirium for Spinal Fusion Patients. J Perianesth Nurs. 2019 Aug;34(4):779-788. doi: 10.1016/j.jopan.2018.11.009. Epub 2019 Feb 10. PMID 30745263
- [Derived] Raymond BL, Allen BFS, Freundlich RE, McEvoy MD, Parrish CG, Ruble SR, Scharfman KH, Wanderer JP, Gao Y, Choi L, Dear ML, Master H, Rice TW, Kertai MD; Vanderbilt Learning Healthcare System Platform Investigators. IMpact of PerioperAtive KeTamine on Enhanced Recovery After abdominal Surgery (IMPAKT ERAS): a pragmatic randomised single-cluster trial. Br J Anaesth. 2025 Dec;135(6):1770-1778. doi: 10.1016/j.bja.2025.08.001. Epub 2025 Sep 3. PMID 40903379
- [Derived] Raymond BL, Allen BFS, Freundlich RE, Parrish CG, Jayaram JE, Wanderer JP, Rice TW, Lindsell CJ, Scharfman KH, Dear ML, Gao Y, Hiser WD, McEvoy MD; Vanderbilt Learning Healthcare System Platform Investigators. The IMpact of PerioperAtive KeTamine on Enhanced Recovery after Abdominal Surgery (IMPAKT ERAS): protocol for a pragmatic, randomized, double-blinded, placebo-controlled trial. BMC Anesthesiol. 2023 Jun 30;23(1):227. doi: 10.1186/s12871-023-02177-y. PMID 37391729
- [Derived] Raymond BL, Allen BFS, Freundlich RE, Parrish CG, Jayaram JE, Wanderer JP, Rice TW, Lindsell CJ, Scharfman KH, Dear ML, Gao Y, Hiser WD, McEvoy MD. The IMpact of PerioperAtive KeTamine on Enhanced Recovery after Abdominal Surgery (IMPAKT ERAS): protocol for a pragmatic, randomized, double-blinded, placebo-controlled trial. Res Sq [Preprint]. 2023 Mar 24:rs.3.rs-2639840. doi: 10.21203/rs.3.rs-2639840/v1. PMID 36993617

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Saline
Started | 798 | 772
Completed | 770 | 752
Not Completed | 28 | 20
Not completed — post randomization exclusion | 28 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Saline | Total
Number analyzed (Participants) | 770 | 752 | 1522
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.9 [46.7 to 69.2] | 57.8 [44.3 to 67.8] | 58.3 [45.3 to 68.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 371 | 380 | 751
  Male | 399 | 372 | 771
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 686 | 660 | 1346
  Black or African American | 58 | 67 | 125
  Asian | 3 | 11 | 14
  Other | 15 | 9 | 24
  Hispanic/Latino | 3 | 3 | 6
  Unknown | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 770 | 752 | 1522
Opioid status [Count of Participants; unit: Participants]
  Exposed | 82 | 76 | 158
  Naive | 688 | 676 | 1364
BMI (kg/m²) [Median (Inter-Quartile Range); unit: kg/m²] | 27.3 [23.7 to 31.3] | 27.6 [23.6 to 32.0] | 27.4 [23.6 to 31.6]

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: The participants length of stay, from anesthesia beginning to discharge, measured in days
Time Frame: From surgery start until discharge, typically 3-5 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 770 | 752
days | 5.0 [4.0 to 8.0] | 5.0 [3.0 to 7.2]

2. Secondary Outcome: Total Consumption of Inpatient Opioids
Description: Inpatient opioid consumption measured in morphine milligram equivalents
Time Frame: From hospital admission until discharge, typically 3-5 days
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 770 | 752
MME | 82.5 [37.5 to 158.0] | 90.0 [45.0 to 158.0]

3. Secondary Outcome: Number of Participants With Ileus
Description: Number of participants reporting ileus requiring gastric decompression as defined by orogastric or nasogastric tube placement in the postoperative period.
Time Frame: From hospital admission until discharge, typically 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 770 | 752
Participants | 71 | 37

4. Secondary Outcome: Number of Participants Who Encounter Rapid Response Team Activation
Description: Number of participants who encounter rapid response team activation within 72 hours post-operation. This is as a binary outcome
Time Frame: From hospital admission until discharge, typically 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 770 | 752
Participants | 39 | 26

5. Secondary Outcome: Number of Participants Who Experienced ICU Transfer
Description: Number of participants who experienced transfer to ICU. This is as a binary outcome
Time Frame: From hospital admission until discharge, typically 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 770 | 752
Participants | 44 | 22

6. Secondary Outcome: Number of Participants Who Experienced Adverse Side Effects
Description: Total number of side effects (hallucination, sedation, lightheadedness, patient request) as adverse reactions requiring early cessation.
Time Frame: From hospital admission until discharge, typically 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 770 | 752
Participants
  Met Early Discharge Milestones | 96 | 130
  Patient Preference for Mild Side Effects | 83 | 39
  Debilitating Hallucinations | 19 | 7
  Debilitating Dizziness | 64 | 11
  Hemodynamic Instability | 12 | 6
  Other Severe Side Effect | 71 | 37

ADVERSE EVENTS:
Time Frame: Monitored from enrollment to time of hospital discharge, approximately 28 days
Arm/Group | Ketamine | Saline
All-Cause Mortality (participants affected / at risk) | 1/770 | 0/752
Serious Adverse Events (participants affected / at risk) | 0/770 | 1/752
Other Adverse Events (participants affected / at risk) | 322/770 | 163/752
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=770) | Saline (N=752)
Fall (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=770) | Saline (N=752)
Patient Preference forMild Side Effects (General disorders) | 83 | 39
Debilitating Hallucinations (Psychiatric disorders) | 19 | 7
Debilitating Dizziness (Nervous system disorders) | 64 | 11
Hemodynamic Instability (Vascular disorders) | 12 | 6
Rapid Response Activation (General disorders) | 39 | 26
Transfer to the ICU (Surgical and medical procedures) | 44 | 22
Ileus Requiring NG Decompression (Gastrointestinal disorders) | 63 | 48 — ileus requiring gastric decompression as defined by orogastric or nasogastric tube placement in the postoperative period
Other Severe Side Effect (General disorders) | 71 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04625283/Prot_001.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT04625283/SAP_002.pdf
  • Informed Consent Form (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT04625283/ICF_000.pdf